CLINICAL TRIAL: NCT07027540
Title: Unilateral Right-Sided Erector Spinae Plane Block for Analgesia in Laparoscopic Cholecystectomy: Does the Volume Matter? A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eithar Mahmoud Abd-Elsalm, Doctor at Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uni Rt ESPB LAB Cholecystectom
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Adult patients will take a total 35 ml of Bupivacaine 0.25% and 2mg of Dexmethasone in the right T7.
  Interventions: Drug: 2mg of dexamethasone; Drug: 35 ml of Bupivacaine 0.25%
- Group B (Active Comparator): Adult patients will take a total 20 ml of Bupivacaine 0.25% and 2mg of dexamethasone in the right T7.
  Interventions: Drug: Bupivacaine 0.25% 20ml; Drug: 2mg of dexamethasone

INTERVENTIONS:
Drug: Bupivacaine 0.25% 20ml — Adult patients will take a total 20 ml of Bupivacaine 0.25%
  Arms: Group B
Drug: 2mg of dexamethasone — 2mg of dexamethasone in the right T7
Drug: 35 ml of Bupivacaine 0.25% — Adult patients will take a total 35 ml of Bupivacaine 0.25%
  Arms: Group A

SUMMARY:
Laparoscopic cholecystectomy is one of the most common surgeries today, cause it has many advantages over open cholecystectomy. (1) Although these advantages pain remains a big problem after laparoscopic cholecystectomy which causes patient admission or readmission. (2) This post-operative laparoscopic cholecystectomy pain causes extreme patient discomfort, extended post-anesthesia care unit stay, and restricts early recovery. (3) To overcome this problem, there were trials of inta abdominal instillation with local anesthetics with no positive results (4,5), so they combined this with local infiltration at the laparoscopic access sites (6,7) with no satisfactory postoperative analgesia. (6,8,9).

With more attention to regional anesthesia as part of multimodal analgesia, different techniques have been used for post-LC pain control, such as paravertebral block (10), rectus sheath block (11), transversus abdominis plane block (12), intercostal nerve block (13), subcostal transversus abdominal plane block (STAP), thoracic epidural, and erector spinae plane block.

Erector spinae plane block which was first described for the treatment of thoracic neuropathic pain, is a peri-paravertebral regional anesthesia technique that has since been reported as an effective technique for the prevention of postoperative pain in various surgeries. (14) Case reports and randomized control trials have shown the efficacy of bilateral ESPB for pain control after LC , though the effects of Unilateral ESPB have not been extensively studied yet. A trial by Poupak Rahimzadeh et al, concluded that a single-shot, right-sided, unilateral ESPB with 20 ml volume LA decreases post-LC opioid consumption and pain The exact mechanism of action of the erector spinae plane (ESP) block remains unclear. Schwartzmann et al. used MRI to investigate this and identified three main mechanisms: spread to the paravertebral space through the intertransverse soft tissue, circumferential epidural spread via the intervertebral foramina, and intercostal spread (15).

The circumferential spread of local anesthetic into the epidural space opens the question of the possibility of contralateral spread, which was discussed by Tulgar et al, a case study that found bilateral sensory block caused by a unilateral ESPB with 30 ml volume of local anesthetic (16).

Based on these findings, we hypothesize that increasing the volume of local anesthetic may enhance the efficacy of the block by promoting wider spread, potentially resulting in improved analgesia and even bilateral sensory blockade following a unilateral injection.

This study aims to answer the question: Can unilateral ESPB with high volume result in superior analgesia for LC and perhaps bilateral block The primary outcome is the numeric rating scale (NRS) score at 12h postoperative

ELIGIBILITY:
Inclusion Criteria:

* Adult patients within age; (18-60)
* Body mass index (BMI); (18-30)
* ASA I - II

Exclusion Criteria:

* Patient refusal to participate in the study Allergy to local anesthetics Coagulopathy Morbid obesity Decreased pulmonary reserve Cardiac disorder Renal dysfunction Pre-existing neurological deficit Psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
NRS score after 12 hours in the 2 groups. | 12 hours
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable